CLINICAL TRIAL: NCT02709369
Title: Functional and Physiological Effects of High-resolution, Relational, Resonance-based, Electroencephalic Mirroring (HIRREM) for Neurological, Cardiovascular and Psychophysiological Disorders
Brief Title: HIRREM Developmental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00017651
Record Dates: First submitted 2016-03-04; First posted 2016-03-16 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2018-11

CONDITIONS: Sleep Initiation and Maintenance Disorders; Anxiety; Post-Traumatic Stress Disorder; Hot Flashes; Headache; Traumatic Brain Injury; Post Concussion Symptoms
Keywords: HIRREM; Neuro-technology; Closed-loop; Acoustic stimulation; Allostatic; heart rate variability; baroreflex sensitivity; traumatic brain injury; sports concussion; PTSD; hot flashes; headache; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic; Hot Flashes; Headache; Brain Injuries, Traumatic; Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Active HIRREM (Experimental): This is a single site, single-arm, open-label, developmental study. Participants are recruited to receive eight to twenty sessions of High-resolution, relational, resonance-based electroencephalic mirroring (HIRREM), in addition to their usual care.
  Interventions: Device: HIRREM

INTERVENTIONS:
Device: HIRREM — HIRREM is a noninvasive, closed-loop, allostatic, acoustic stimulation neuro-technology to facilitate recipient-unique relaxation, auto-calibration, and self-optimization of cortical neural oscillations by reflecting auditory tones in near real time. After an initial HIRREM assessment, evaluating patterns of brain electrical rhythms, subjects get a series of 90-120 minute HIRREM sessions, including 5 to 9 individualized protocols. A protocol is a combination of sensor montage and specific software design, during which dominant brain frequencies, recorded at high spectral resolutions, are translated to audible tones, and reflected back via earphones with as little as 8 milliseconds delay. Protocols are received sitting or reclining in a chair, some with eyes open, others eyes closed.

SUMMARY:
The purpose of this study is to explore the functional and physiological effects associated with the use of High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM), as supplemental care, for symptoms of neurological, cardiovascular, and neuropsychological disorders. This is a non-randomized, open label, and unblinded before-and-after trial, evaluating the effect of HIRREM on an objective, physiological common denominator (heart rate variability, HRV), across a variety of relevant conditions, as well as changes in clinical symptoms inventories, to generate hypotheses and pilot data for investigation in future proposals.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults and children aged 11 years and older.
* Subjects who are over the age of 18 must be able to give informed consent. Children must be able to sign an assent form and have a signed parental permission form.
* Subjects must have the ability to comply with basic instructions and be able to sit still comfortably with the sensor leads attached.
* Subjects previously diagnosed with a neurologic, cardiovascular, or psychophysiological disease such as attention deficit hyperactivity disorder, Asperger Syndrome, chronic pain, dyslexia, depression, insomnia, migraines, anxiety, PTSD, substance abuse disorder, traumatic brain injury, and others.

Exclusion Criteria:

* Subjects who fail to meet inclusion criteria.
* Subjects who are unable, unwilling, or incompetent to provide informed consent, assent and/or parental permission.
* Subjects physically unable to come to the study visits.
* Subjects with a known seizure disorder.
* Subjects with severe bilateral hearing impairment (HIRREM requires the use of headphones).
* Subjects receiving ongoing treatment with opiate, benzodiazepine, anti-psychotic or sleep medications, as well as some anti-depressants or stimulants, except those cases deemed acceptable by the principal investigator.
* Subjects with anticipated and ongoing use of recreational drugs except when deemed acceptable by the principal investigator.

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-08-23 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H Tegeler, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Department of Neurology, Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared in publications and presentations. No plan to formally make individual participant data available for this exploratory study

REFERENCES:
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Background] Tegeler CH, Kumar SR, Conklin D, Lee SW, Gerdes L, Turner DP, Tegeler CL, C Fidali B, Houle TT. Open label, randomized, crossover pilot trial of high-resolution, relational, resonance-based, electroencephalic mirroring to relieve insomnia. Brain Behav. 2012 Nov;2(6):814-24. doi: 10.1002/brb3.101. Epub 2012 Oct 28. PMID 23170244
- [Background] Tegeler CH, Lee SW, Shaltout HA. Significance of right anterior insula activity for mental health intervention. JAMA Psychiatry. 2014 Mar;71(3):336. doi: 10.1001/jamapsychiatry.2013.3507. No abstract available. PMID 24599239
- [Background] Gerdes L, Tegeler CH, Lee SW. A groundwork for allostatic neuro-education. Front Psychol. 2015 Aug 17;6:1224. doi: 10.3389/fpsyg.2015.01224. eCollection 2015. PMID 26347688
- [Result] Lee SW, Gerdes L, Tegeler CL, Shaltout HA, Tegeler CH. A bihemispheric autonomic model for traumatic stress effects on health and behavior. Front Psychol. 2014 Aug 1;5:843. doi: 10.3389/fpsyg.2014.00843. eCollection 2014. PMID 25136325
- [Result] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Pajewski NM. Reduction in menopause-related symptoms associated with use of a noninvasive neurotechnology for autocalibration of neural oscillations. Menopause. 2015 Jun;22(6):650-5. doi: 10.1097/GME.0000000000000422. PMID 25668305
- [Result] Tegeler CH, Shaltout HA, Tegeler CL, Gerdes L, Lee SW. Rightward dominance in temporal high-frequency electrical asymmetry corresponds to higher resting heart rate and lower baroreflex sensitivity in a heterogeneous population. Brain Behav. 2015 Jun;5(6):e00343. doi: 10.1002/brb3.343. Epub 2015 May 1. PMID 26085968
- [Result] Fortunato JE, Tegeler CL, Gerdes L, Lee SW, Pajewski NM, Franco ME, Cook JF, Shaltout HA, Tegeler CH. Use of an allostatic neurotechnology by adolescents with postural orthostatic tachycardia syndrome (POTS) is associated with improvements in heart rate variability and changes in temporal lobe electrical activity. Exp Brain Res. 2016 Mar;234(3):791-8. doi: 10.1007/s00221-015-4499-y. Epub 2015 Dec 8. PMID 26645307
- [Result] Tegeler CH, Tegeler CL, Cook JF, Lee SW, Gerdes L, Shaltout HA, Miles CM, Simpson SL. A Preliminary Study of the Effectiveness of an Allostatic, Closed-Loop, Acoustic Stimulation Neurotechnology in the Treatment of Athletes with Persisting Post-concussion Symptoms. Sports Med Open. 2016 Dec;2(1):39. doi: 10.1186/s40798-016-0063-y. Epub 2016 Sep 14. PMID 27747793
- [Derived] Tegeler CH, Cook JF, Tegeler CL, Hirsch JR, Shaltout HA, Simpson SL, Fidali BC, Gerdes L, Lee SW. Clinical, hemispheric, and autonomic changes associated with use of closed-loop, allostatic neurotechnology by a case series of individuals with self-reported symptoms of post-traumatic stress. BMC Psychiatry. 2017 Apr 19;17(1):141. doi: 10.1186/s12888-017-1299-x. PMID 28420362

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active HIRREM
Started | 300
Completed | 273
Not Completed | 27
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 10
Not completed — Did not received intervention | 2

BASELINE CHARACTERISTICS:
Arm/Group | Active HIRREM
Number analyzed (Participants) | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 228
  >=65 years | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 15
  Asian | 5
  Hispanic or Latino | 3
  White | 276
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 300

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Variability Standard Deviation of NN Intervals (SDNN)
Description: Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval
Time Frame: Baseline/Enrollment visit
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
milliseconds | 44.41 (22.94)

2. Primary Outcome: Heart Rate Variability (SDNN)
Description: Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval
Time Frame: Up to 2 weeks after the intervention is completed
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
milliseconds | 54.82 (30.63)

3. Primary Outcome: Baroreflex Sensitivity High Frequency (HF) Alpha
Description: Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis using Nevrokard Baroreflex Sensitivity (BRS) software.
Time Frame: Baseline/Enrollment visit
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms^2 | 18.81 (14.45)

4. Primary Outcome: Baroreflex Sensitivity High Frequency (HF) Alpha
Description: as for outcome 3
Time Frame: Up to two weeks after the intervention is completed
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms^2 | 26.68 (20.69)

5. Primary Outcome: Baroreflex Sensitivity Sequence Up
Description: as for outcome 3
Time Frame: Baseline/Enrollment visit
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 226
ms/mmHg | 15.39 (13.88)

6. Primary Outcome: Baroreflex Sensitivity Sequence Up
Description: as for outcome 3
Time Frame: Up to two weeks after the intervention is completed
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 226
ms/mmHg | 14.15 (11.56)

7. Primary Outcome: Baroreflex Sensitivity Sequence Down
Description: as for outcome 3
Time Frame: Baseline/Enrollment visit
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms/mmHg | 14.15 (11.56)

8. Primary Outcome: Baroreflex Sensitivity Sequence Down
Description: as for outcome 3
Time Frame: Up to two weeks after the intervention is completed
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms/mmHg | 20.73 (16.76)

9. Primary Outcome: Baroreflex Sensitivity Sequence All
Description: as for outcome 3
Time Frame: Baseline/Enrollment visit
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms/mmHg | 14.63 (11.80)

10. Primary Outcome: Baroreflex Sensitivity Sequence All
Description: as for outcome 3
Time Frame: Up to 2 weeks after the intervention is completed
Population: BIOPAC device was acquired prior to subject 38. Other entries were excluded due to missing or dropped heartbeats.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Arm/Group | Active HIRREM
Number analyzed (Participants) | 227
ms/mmHg | 20.74 (16.30)

11. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D is a 20-item survey assessing affective depressive symptomatology to screen for risk of depression. Scores range from 0-60, with a score of 16 commonly used as a clinically relevant cut-off. Higher scores suggest the presence of more symptomatology.
Time Frame: enrollment visit/baseline
Population: CES-D was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 233
score on a scale | 18.12 (12.16)

12. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: as for outcome 11
Time Frame: 1-2 weeks after intervention is completed
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 233
score on a scale | 10.00 (8.96)

13. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Description: as for outcome 11
Time Frame: 4-8 weeks after completion of the intervention
Population: CES-D was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 115
score on a scale | 8.91 (8.28)

14. Secondary Outcome: Euro Quality of Life--Five Dimension (EQ-5D)
Description: The EQ-5D is a brief, standardized measure of health status developed by the EuroQol Group, and is a paper and pencil survey providing a single index value for health status. The score reported is current health status which ranges from 0 to 100 with a higher score denoting a better outcome.
Time Frame: enrollment visit/baseline
Population: EQ-5D was added as a study measure at subject 79. Entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 202
score on a scale | 69.55 (19.69)

15. Secondary Outcome: Euro Quality of Life--Five Dimension (EQ-5D)
Description: as for outcome 14
Time Frame: 1-2 weeks after the intervention is completed
Population: EQ-5D was added as a study measure at subject 79. Entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 202
score on a scale | 79.12 (16.42)

16. Secondary Outcome: Euro Quality of Life--Five Dimension (EQ-5D)
Description: as for outcome 14
Time Frame: 4-8 weeks after completion of the intervention
Population: EQ-5D was added as a study measure at subject 79. Entries were excluded if there was incomplete or missing data. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 151
score on a scale | 78.36 (17.84)

17. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: The Generalized Anxiety Disorder-7 (GAD-7) is a seven item screening tool for anxiety that is widely used in primary care. Scores range from 0 to 21 with higher scores suggesting anxiety.
Time Frame: enrollment visit/baseline
Population: GAD-7 was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 167
score on a scale | 8.31 (6.01)

18. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: as for outcome 17
Time Frame: 1-2 weeks after the intervention is completed
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 167
score on a scale | 4.35 (4.19)

19. Secondary Outcome: Generalized Anxiety Disorder-7 (GAD-7)
Description: as for outcome 17
Time Frame: 4-8 weeks after completion of the intervention
Population: GAD-7 was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 133
score on a scale | 3.66 (3.49)

20. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI measures the severity of insomnia symptoms. The ISI is a 7 question measure, with responses from 0-4 for each question, yielding scores ranging from 0-28 where lower scores denote a healthier sleep quality.
Time Frame: enrollment visit/baseline
Population: Entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 272
score on a scale | 13.47 (7.17)

21. Secondary Outcome: Insomnia Severity Index (ISI)
Description: as for outcome 20
Time Frame: 1-2 weeks after the intervention is completed
Population: Entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 270
score on a scale | 7.09 (5.90)

22. Secondary Outcome: Insomnia Severity Index (ISI)
Description: as for outcome 20
Time Frame: 4-8 weeks after completion of the intervention
Population: Entries were excluded if there was incomplete or missing data. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 160
score on a scale | 6.22 (5.43)

23. Secondary Outcome: Posttraumatic Stress Disorder Checklist (PCL-C)
Description: The PCL - Civilian (C) is a symptom checklist to measure stress severity due to a traumatic experience, in civilian settings. Seventeen items are rated on a Likert scale with a composite score range of 17 to 85. A score of 44 or higher correlates with probability of civilian-related PTSD.
Time Frame: enrollment visit/baseline
Population: Entries were excluded if there was incomplete or missing data. Scale was exploratory and only administered to people who self-reported trauma or PTSD on medical history form.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 179
score on a scale | 38.75 (15.43)

24. Secondary Outcome: Posttraumatic Stress Disorder Checklist (PCL)
Description: as for outcome 23
Time Frame: 1-2 weeks after the intervention is completed
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 179
score on a scale | 28.50 (11.37)

25. Secondary Outcome: Posttraumatic Stress Disorder Checklist (PCL)
Description: as for outcome 23
Time Frame: 4-8 weeks after completion of the intervention
Population: Entries were excluded if there was incomplete or missing data. Scale was exploratory and only administered to people who self-reported trauma or PTSD on medical history form. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 91
score on a scale | 26.13 (9.58)

26. Secondary Outcome: Rivermead Post-Concussion Symptoms Questionnaire (RPQ)
Description: The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is a 16-item survey that assesses the severity of the most common post-concussion symptoms on a scale of 0 to 4, with a total score range from 0 to 64 with 64 denoting the greatest symptom severity.
Time Frame: enrollment visit/baseline
Population: Entries were excluded if there was incomplete or missing data. Scale was exploratory and only administered to people who self-reported TBI or concussion on medical history form.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 48
score on a scale | 29.60 (12.82)

27. Secondary Outcome: Rivermead Post-Concussion Symptoms Questionnaire (RPQ)
Description: The Rivermead Post-Concussion Symptoms Questionnaire (RPQ) is a 16-item survey that assesses the severity of the most common post-concussion symptoms on a scale of 0 to 4, with a total score range from 0 to 64 with a higher score denoting the greatest symptom severity.
Time Frame: 1-2 weeks after the intervention is completed
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 48
score on a scale | 15.79 (13.96)

28. Secondary Outcome: Rivermead Post-Concussion Symptoms Questionnaire (RPQ)
Description: as for outcome 26
Time Frame: 4-8 weeks after completion of the intervention
Population: Entries were excluded if there was incomplete or missing data. Scale was exploratory and only administered to people who self-reported TBI or concussion on medical history form. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active HIRREM
Number analyzed (Participants) | 35
score on a scale | 16.89 (14.74)

29. Secondary Outcome: Drop Stick Reaction Testing
Description: Reaction testing is measured by a drop-stick apparatus that has been validated as a way to quantify the impact of athletic concussion on psychomotor performance. Following two practice trials, participants perform eight trials, and a mean distance value is calculated. Better reaction time is denoted by a lower score. The scores range from 0 to 100.
Time Frame: enrollment visit/baseline
Population: Drop stick reaction testing was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Active HIRREM
Number analyzed (Participants) | 213
cm | 27.20 (8.25)

30. Secondary Outcome: Drop Stick Reaction Testing
Description: as for outcome 29
Time Frame: 1-2 weeks after the intervention is completed
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Active HIRREM
Number analyzed (Participants) | 213
cm | 23.40 (6.78)

31. Secondary Outcome: Drop Stick Reaction Testing
Description: as for outcome 29
Time Frame: 4-8 weeks after completion of the intervention
Population: Drop stick reaction testing was temporarily removed as approved measure of depression (35 subjects). Other entries were excluded if there was incomplete or missing data. Late data collection visit was added at after participant 65. Out of town subjects typically were not able to make it back for late data collections.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Active HIRREM
Number analyzed (Participants) | 90
cm | 22.58 (5.78)

32. Other Pre Specified Outcome: Heart Rate Variability Standard Deviation of NN Intervals (SDNN)
Description: Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval
Time Frame: 4-8 weeks after completion of the intervention
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Baroreflex Sensitivity High Frequency (HF) Alpha
Description: as for outcome 3
Time Frame: 4-8 weeks after completion of the intervention
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Baroreflex Sensitivity Sequence Up
Description: as for outcome 3
Time Frame: 4-8 weeks after completion of the intervention
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Baroreflex Sensitivity Sequence Down
Description: as for outcome 3
Time Frame: 4-8 weeks after completion of the intervention
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Baroreflex Sensitivity Sequence All
Description: as for outcome 3
Time Frame: 4-8 weeks after completion of the intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Informed consent until 4-8 weeks after completion of the intervention
Arm/Group | Active HIRREM
All-Cause Mortality (participants affected / at risk) | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT02709369/Prot_SAP_000.pdf